CLINICAL TRIAL: NCT00023920
Title: A Phase II Study of Bevacizumab (rhuMab VEGF, NSC 704865), Idarubicin and Cytarabine in Patients With Chronic Myeloid Leukemia in Blast Phase
Brief Title: Bevacizumab, Idarubicin, and Cytarabine in Treating Patients With Blast Phase Chronic Myelogenous Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02405; ID00-323; N01CM17003 (NIH); CDR0000068876 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Blastic Phase Chronic Myelogenous Leukemia; Chronic Myelogenous Leukemia, BCR-ABL1 Positive
MeSH Terms: conditions — Blast Crisis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Bevacizumab; Idarubicin; Cytarabine

ARMS (1):
- Treatment (bevacizumab, idarubicin, cytarabine) (Experimental): Patients receive bevacizumab IV over 90 minutes once on day -13. Patients then receive bevacizumab IV over 90 minutes and idarubicin IV on days 1 and 15 and cytarabine subcutaneously (SC) once daily beginning on day 1. Treatment repeats every 4 weeks for a maximum of 3 courses. Patients with responding disease receive maintenance therapy comprising bevacizumab IV over 90 minutes on days 1 and 15, idarubicin IV on day 1, and cytarabine SC once daily beginning on day 1. Treatment repeats every 4 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Drug: idarubicin; Drug: cytarabine

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Drug: idarubicin — Given IV
  Other Names: 4-demethoxydaunorubicin; 4-DMDR; DMDR; IDA
Drug: cytarabine — Given SC
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside

SUMMARY:
This phase II trial is to see if combining bevacizumab with idarubicin and cytarabine works better in treating patients who have blast phase chronic myelogenous leukemia. Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or deliver cancer-killing substances to them. Drugs used in chemotherapy, such as idarubicin and cytarabine, work in different ways to stop cancer cells from dividing so they stop growing or die. Combining monoclonal antibody therapy with chemotherapy may be an effective treatment for blast phase chronic myelogenous leukemia

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the anti-leukemic activity of bevacizumab, idarubicin, and cytarabine in patients with blastic phase chronic myelogenous leukemia.

II. Determine the toxicity profile of this regimen in these patients. III. Determine the effect of bevacizumab on angiogenesis in these patients.

OUTLINE:

Patients receive bevacizumab IV over 90 minutes once on day -13. Patients then receive bevacizumab IV over 90 minutes and idarubicin IV on days 1 and 15 and cytarabine subcutaneously (SC) once daily beginning on day 1. Treatment repeats every 4 weeks for a maximum of 3 courses. Patients with responding disease receive maintenance therapy comprising bevacizumab IV over 90 minutes on days 1 and 15, idarubicin IV on day 1, and cytarabine SC once daily beginning on day 1. Treatment repeats every 4 weeks for 2 years in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Philadelphia chromosome-positive blastic phase chronic myelogenous leukemia (CML), defined by 1 of the following:

  * At least 30% blasts in peripheral blood and/or bone marrow
  * Presence of extramedullary disease
* Performance status - Zubrod 0-2
* At least 8 weeks
* No prior coagulopathies
* Bilirubin no greater than 1.5 mg/dL
* INR less than 2
* PTT no greater than 60 seconds
* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min
* No nephrotic syndrome
* No uncontrolled hypertension
* No New York Heart Association class II-IV heart disease
* No prior thrombotic events
* LVEF ≥ 50%
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No more than 2 prior chemotherapy regimens (no more than 1 regimen containing cytarabine) for CML in blast crisis
* Prior hydroxyurea allowed
* Prior imatinib mesylate allowed
* At least 10 days since prior anticoagulants
* No concurrent anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2001-07; Primary Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Improvement in response rate | Up to 3 years
Controlled toxicity rate graded according to NCI Common Toxicity Criteria | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States